CLINICAL TRIAL: NCT04675970
Title: Long Term Follow up Patients With Premature Ovarian Failure ex Vivo Gene Therapy Using Autologous Mesenchymal Stem Cell and Mesenchymal Stem Cell Lyophilisate
Brief Title: Long Term Follow up Patients With Premature Ovarian Failure ex Vivo Gene Therapy
Acronym: UB-OVF
Status: Completed | Type: Observational
Sponsor: Ukraine Association of Biobank (Other)
Responsible Party: Sponsor
Other Study IDs: UAB1220-2
Record Dates: First submitted 2020-12-13; First posted 2020-12-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Primary Ovarian Insufficiency; Premature Ovarian Failure
Keywords: Premature ovarian failure; stem cell therapy; mesenchymal stem cell
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Product in a Institute of Bio-Stem Cell rehabilitation UAB - sponsored clinical trial who agree to participate in this study

SUMMARY:
This is a multi-centers of long term safety and efficacy follow up study for patients with premature ovarian failure (the women aged younger than 40 years, who present with amenorrhoea, hypergonadotropic hypogonadism, and infertility) who have been treated with ex vivo gene therapy drug product in Institute of Bio-Stem Cell Rehabilitation UAB - sponsored clinical studies. After completing the parent clinical study (approximately 6 month), eligible subject will be followed for additional 2 years for total of 2 years and 6 month post drug product infusion. No investigation drug product will be administered in the study

ELIGIBILITY:
Inclusion Criteria:

Provision of written informed consent for this study by subjects or as applicable parent legal guardian. Treated with drug product for therapy of premature ovarian insufficiency in a Institute Bio-Stem Cell Rehabilitation UAB clinical study.

Diagnosed of premature ovarian insufficiency ESHRE:

* Women age of 18 to 40 years
* Have experienced 4 months of oligo/amenorrhea
* Two serum follicle-stimulating hormone (FSH was >40 mIU/ml levels in the menopausal range, obtained at least a month apart
* lower FSH levels ( 25 mIU/ml)
* anti-Müllerian hormone (AMH) serum levels ( 3.0 ng/ml)

Exclusion Criteria:

There are no exclusion criteria for this study

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Patients with premature ovarian insufficiency (Diagnostic criteria of ESHRE) who have been treated with ex vivo gene therapy product in a Institute Bio-Stem Cell Rehabilitation UAB clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Antral follicular count (AFC) serum levels | 2 years
  Antral follicular count (AFC) <5-7 follicles
anti-Müllerian hormone (AMH) serum levels | 2 years
  AMH <0.5-1.1 ng/ml

SECONDARY OUTCOMES:
Regular menstruation and/or pregnancy | 2 years
  regular menstruation for 5 months and\or pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Bio-Stem Cell Rehabilitation, Kharkiv, Ukraine